CLINICAL TRIAL: NCT02307591
Title: Clinical Study to Assess Efficacy and Safety of Amiodarone in Treating Patients With Ebola.
Brief Title: Clinical Study to Assess Efficacy and Safety of Amiodarone in Treating Patients With Ebola. Virus Disease (EVD) in Sierra Leone. EASE (EMERGENCY Amiodarone Study Against Ebola)
Acronym: EASE
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The Study could not be started due to an insufficient number of new EVD cases.
Sponsor: Emergency NGO Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EASE
Record Dates: First submitted 2014-11-21; First posted 2014-12-04 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best Supportive Care (Active Comparator): Dehydration Ringer's lactate solution or normal saline intravenously Electrolytes should be monitored at regular intervals and corrected as long as vomiting and/or diarrhoea persist Fever intravenous Paracetamol Antimicrobial treatment Prophylactic 5-days course with Ampicillin should be used Pain Paracetamol,Tramadol or Pentazocine Central nervous system disturbances If a patient is restless or confused, prescribe a light sedation utilizing Midazolam, Propofol or Ketamine, preferably in association with Diazepam or Midazolam Seizures Diazepam Vomiting antiemetic medications may provide some relief and facilitate the rehydration Dyspepsia in adults, Omeprazole Diarrhoea in adults, Loperamide Acute bleeding leading to signs of haemorrhagic shock should be treated with whole blood transfusion and supportive care. Patients haemodynamically stable should not be transfused if the Hb level is >7 mg% Septic shock intensive support care Malaria in case of positive initial test, Artesunate
  Interventions: Drug: Best Supportive Care
- Best Supportive Care + Amiodarone (Experimental): This treatment will be provided to patients in the experimental arm only in addition to best supportive care scheme .
  During the first 3 days of treatment, the drug must be administered in Glucose 5% solution. Deliver through the largest possible vein inserting a long catheter (if possible a CVP line).
  Day 1. Dose: 20 mg/kg/die i.v. deliver a loading dose of 5mg/kg in the 1st hour, followed by continuous infusion during the remaining 23 hours.
  Example: 20 mg /kg of Amiodarone in 500 cc of Glucose 5%. Deliver 125 ml during the 1st hour followed by 16 ml/hour for the remaining 23 hours.
  Day 2 - Day 3. Dose: 20 mg/kg/die i.v. Continuous infusion over 24 hrs. Example: Glucose 5% 500 ml containing 20 mg/kg of Amiodarone (infusion speed = 21 ml/hour).
  Day 4 to Day 10. If no significant diarrhea and/or vomiting, shift to oral intake of Amiodarone as follows:
  * Adults: 200 mg tablets, 3 times a day, according to the body weight (30mg/Kg)
  * Children < 29 kg: 5 mg/kg 3 times a day
  Interventions: Drug: Best Supportive Care + Amiodarone

INTERVENTIONS:
Drug: Best Supportive Care — Dehydration Ringer's lactate solution or normal saline intravenously Electrolytes should be monitored at regular intervals and corrected as long as vomiting and/or diarrhoea persist Fever intravenous Paracetamol Antimicrobial treatment Prophylactic 5-days course with Ampicillin should be used Pain Paracetamol,Tramadol or Pentazocine Central nervous system disturbances If a patient is restless or confused, prescribe a light sedation utilizing Midazolam, Propofol or Ketamine, preferably in association with Diazepam or Midazolam Seizures Diazepam Vomiting antiemetic medications may provide some relief and facilitate the rehydration Dyspepsia in adults, Omeprazole Diarrhoea in adults, Loperamide Acute bleeding leading to signs of haemorrhagic shock should be treated with whole blood transfusion and supportive care. Patients haemodynamically stable should not be transfused if the Hb level is >7 mg% Septic shock intensive support care Malaria in case of positive initial test, Artesunate
  Arms: Best Supportive Care
Drug: Best Supportive Care + Amiodarone — This treatment will be provided to patients in the experimental arm only in addition to best supportive care scheme .
  During the first 3 days of treatment, the drug must be administered in Glucose 5% solution. Deliver through the largest possible vein inserting a long catheter (if possible a CVP line).
  Day 1. Dose: 20 mg/kg/die i.v. deliver a loading dose of 5mg/kg in the 1st hour, followed by continuous infusion during the remaining 23 hours.
  Example: 20 mg /kg of Amiodarone in 500 cc of Glucose 5%. Deliver 125 ml during the 1st hour followed by 16 ml/hour for the remaining 23 hours.
  Day 2 - Day 3. Dose: 20 mg/kg/die i.v. Continuous infusion over 24 hrs. Example: Glucose 5% 500 ml containing 20 mg/kg of Amiodarone (infusion speed = 21 ml/hour).
  Day 4 to Day 10. If no significant diarrhea and/or vomiting, shift to oral intake of Amiodarone as follows:
  * Adults: 200 mg tablets, 3 times a day, according to the body weight (30mg/Kg)
  * Children < 29 kg: 5 mg/kg 3 times a day
  Arms: Best Supportive Care + Amiodarone

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of amiodarone in the treatment of patients afflicted with Ebola virus disease.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted to the Emergency ETC at Goderich with a clinical diagnosis of Ebola virus disease;
* patient who consent to participate in the study.

Exclusion Criteria:

* negative RT-PCR tests for Ebola virus
* age <2 years
* state of shock upon admission
* onset of fever for more than 6 days
* Glasgow Coma Scale <12
* known contraindications to administration of amiodarone
* positive for HIV antibodies.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 10 days

SECONDARY OUTCOMES:
Adverse events | Day 1-10 , 14
Viral load | Day 2, 5, 10 and 14
Lymphocyte count | Day 2, 5, 10 and 14
IgM anti-Ebola virus antibody titer | Day 2, 5, 10 and 14
IgG anti-Ebola virus antibody titer | Day 2, 5, 10 and 14
Serum concentration of amiodarone | Day 2, 5, 10 and 14
Vital status | Day 14 and 30